CLINICAL TRIAL: NCT00218114
Title: Parallel Groups Study of Divalproex Sodium (Depakote) for Irritable, Explosive Adults & Adolescents
Brief Title: Divalproex Sodium (Depakote) for Explosive Tempers in Adolescents and Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: #4767R; R01DA012234 (NIH)
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Attention Deficit and Disruptive Behavior Disorders; Marijuana Abuse
Keywords: ADHD, disruptive behavior disorder, marijuana abuse
MeSH Terms: conditions — Attention Deficit and Disruptive Behavior Disorders; Marijuana Abuse; Attention Deficit Disorder with Hyperactivity | interventions — Valproic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Divalproex sodium (Depakote). This is a parallel groups design lasting a total of six weeks. Participants will be on a fixed-flexible dosing schedule. The dose of depakote will be raised to 750mgs or 1000mgs, depending on weight, in two weeks to achieve blood levels between 50-130 micrograms per milliliter. If a patient does not achieve this blood level on 750mgs or 1000 mgs, the dose may be raised during the second week.
  Interventions: Drug: Divalproex Sodium
- 2 (Placebo Comparator): This is a parallel groups design lasting a total of six weeks. Participants will be on matching placebo for 250 mgs divalproex sodium (Depakote).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Divalproex Sodium — Participants are titrated over 2 weeks, as tolerated to 10 mgs / pound, and blood levels are checked to determine that the blood level is between 50-110 micrograms / ml.
  Other Names: Depakote
  Arms: 1
Drug: Placebo — Participants will be on matching placebo.
  Arms: 2

SUMMARY:
The purpose of this study is to compare the effectiveness of divalproex sodium (Depakote) versus placebo in treating disruptive behavior disorder and explosive tempers in adolescents and adults.

DETAILED DESCRIPTION:
Disruptive behavior disorders among children and adolescents are readily diagnosed; however, few individuals with such disorders receive drug treatment. Depakote is a mood stabilizing medication that may be beneficial in treating individuals with disruptive behavior disorders. The purpose of this study is to examine the effectiveness of Depakote in reducing temper outbursts and improving mood in individuals with disruptive behavior disorders. In addition, this study will determine the safety and effectiveness of Depakote in treating individuals with substance disorders who also have disruptive behavior disorders.

This study will last 6 weeks. Participants will be randomly assigned to receive treatment with Depakote or placebo. Medication will be given in a single evening dose if tolerated; otherwise, medication will be given twice per day. Participants will be assigned to a fixed-flexible dosing schedule and dosages will increase based on weight. All participants will attend weekly psychotherapy and family counseling sessions throughout the study. Participants who are substance abusers will also receive substance abuse counseling. Weekly study visits will include a physical exam, blood collection, and drug tests. Teachers and guidance counselors will be contacted to assess the participant's behavior from week to week. Some participants will complete a follow-up study, in which they will take part in phone interviews.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for a disruptive behavior disorder (e.g., oppositional/defiant disorder, conduct disorder)
* Explosive temper, defined as four or more outbursts of rage, property destruction, or fighting per month
* Mood liability, defined as having multiple, daily, distinct shifts from normal to irritable mood with withdrawn or boisterous behavior
* Chronic symptoms, defined of at least 1 year duration when not receiving treatment
* Impairment from the above symptoms in two or more areas, including school, the law, family, substance use, peers, or work (as manifested by a GAF score of 55 or less)
* Symptoms not limited to a particular place or to particular intimate relationships
* General good health
* Custodial parent or guardian gives informed consent

Exclusion Criteria:

* History of non drug-induced psychosis
* Seizure or other neurologic disturbance
* Pregnant
* Moderate to severe mental retardation
* Sexually active females who refuse to use an adequate method of contraception for the duration of the study
* Significant medical problems
* Current suicidal or homicidal ideation
* Uses barbiturates
* Refusal to permit weekly contact with school officials
* Bipolar I or II disorder
* Major depressive disorder
* First degree relative with bipolar I or II disorder
* Attention deficit/hyperactivity disorder
* Post traumatic stress disorder
* Clinical evidence of hyperandrogenism in a female
* Liver disease
* Thrombocytopenia
* Pancreatic disease

Ages: 12 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2000-02 (Actual); Primary Completion 2005-02-18 (Actual); Study Completion 2005-02-18 (Actual)

PRIMARY OUTCOMES:
Symptoms of disruptive behavior disorder | 6 weeks
  Measure symptoms of disruptive behavior disorder with the modified overt aggression scale throughout the study and at Week 6

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Donovan, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States